CLINICAL TRIAL: NCT04738877
Title: FEIDIPIDIS Study: Cardiovascular Effects of Marathon Running
Brief Title: Cardiovascular Effects of Marathon Running
Acronym: FEIDIPIDIS
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Evangelia Kouidi, Professor of Sports Medicine, Aristotle University Of Thessaloniki
Other Study IDs: EC-3/2020
Record Dates: First submitted 2021-01-27; First posted 2021-02-04 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Athletes Heart
MeSH Terms: interventions — Exercise Test; Echocardiography; Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Body fat measurement — Body fat measurement using skinfolds
Diagnostic Test: Cardiopulmonary exercise testing — Electrocardiographic exercise testing with ergospirometer on a treadmill
Diagnostic Test: Echocardiography — Transthoracic echocardiography
Diagnostic Test: Blood test — Blood test for measurement of haemoglobin, serum electrolytes, iron, ferritin and vitamins

SUMMARY:
The aim of this study is the investigation of acute cardiovascular responses of marathon runners after the completion of a marathon race (42.2 km), as well as of the determinants of these changes.

ELIGIBILITY:
Inclusion Criteria:

* Marathon runner

Exclusion Criteria:

* Chronic disease, Drugs

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Marathon runners aiming to paricipate in a marathon running race
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Baseline left ventricular (LV) systolic function | Evaluation of athletes within 3 weeks before the marathon running race.
  Evaluation of LV ejection fraction
Baseline LV diastolic function | Evaluation of athletes within 3 weeks before the marathon running race.
  Evaluation of LV filling pressures
Baseline basal right ventricular (RV) function | Evaluation of athletes within 3 weeks before the marathon running race.
  Evaluation of tricuspid annular plane systolic excursion (TAPSE)
Baseline global RV function | Evaluation of athletes within 3 weeks before the marathon running race.
  Evaluation of RV fractional are change (RVFAC)
Post-exercise LV systolic function | Evaluation of athletes immediately after the completion of the marathon running race.
  Evaluation of LV ejection fraction
Post-exercise LV diastolic function | Evaluation of athletes immediately after the completion of the marathon running race.
  Evaluation of LV filling pressures
Post-exercise basal RV function | Evaluation of athletes immediately after the completion of the marathon running race.
  Evaluation of TAPSE
Post-exercise global RV function | Evaluation of athletes immediately after the completion of the marathon running race.
  Evaluation of RVFAC

CONTACTS AND LOCATIONS:
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Greece

REFERENCES:
- [Derived] Christou GA, Pagourelias ED, Deligiannis AP, Kouidi EJ. Exploring the Anthropometric, Cardiorespiratory, and Haematological Determinants of Marathon Performance. Front Physiol. 2021 Sep 3;12:693733. doi: 10.3389/fphys.2021.693733. eCollection 2021. PMID 34539429